CLINICAL TRIAL: NCT05761366
Title: Application of 18F-PSMA PET / CT Imaging in Prostate Specific Membrane Antigen Positive Tumor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCC3688
Record Dates: First submitted 2023-02-19; First posted 2023-03-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Malignancy
Keywords: Malignancy; Prostate Specific Membrane Antigen Positive Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Al18F-PSMA-BCH PET/CT (Experimental): Al18F-PSMA-BCH PET/CT will be performed on patients with suspected or clearly diagnosed PSMA positive-expressing tumors.（including prostate cancer, transitional epithelial carcinoma, colon carcinoma, adenoid cystadenocarcinoma, mesothelioma, hepatocellular carcinoma, cholangiocellular carcinoma, multiple myeloma, etc.）
  Interventions: Drug: Al18F-PSMA-BCH PET/CT

INTERVENTIONS:
Drug: Al18F-PSMA-BCH PET/CT — Patients will be intravenously injected with Al18F-PSMA-BCH and undergo PET/CT scan.
  Other Names: 18F-Thretide PET/CT

SUMMARY:
In this study, Al18F-PSMA-BCH PET/CT will be performed in patients with prostate specific membrane antigen positive tumor, to evaluate the tumour detection efficacy of Al18F-PSMA-BCH PET/CT.

DETAILED DESCRIPTION:
Al18F-PSMA-BCH PET/CT will be performed on patients with suspected or clearly diagnosed PSMA positive-expressing tumors (including prostate cancer, transitional epithelial carcinoma, colon carcinoma, adenoid cystadenocarcinoma, mesothelioma, hepatocellular carcinoma, cholangiocellular carcinoma, multiple myeloma, etc.) , to evaluate the tumour detection efficacy of Al18F-PSMA-BCH PET/CT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected or clearly diagnosed PSMA positive-expressing tumors, including prostate cancer, transitional epithelial carcinoma, colon carcinoma, adenoid cystadenocarcinoma, mesothelioma, hepatocellular carcinoma, cholangiocellular carcinoma, multiple myeloma, etc.
2. Age is 18 or older; No gender limitation.
3. Signed the informed consent.
4. Willing and able to cooperate with all projects in this study.

Exclusion Criteria:

1. Patients with serious neurological diseases,or gastrointestinal tract disease, cardiovascular disease, liver disease, kidney disease, blood system disease, endocrine system disease, respiratory system disease, immune deficiency disease, etc
2. Claustrophobia.
3. Pregnant or lactation women.
4. Received experimental drug or device within 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-10-13 (Estimated); Study Completion 2025-10-13 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of 18F-PSMA PET / CT for the diagnosis of Prostate Specific Membrane Antigen Positive Tumor

CONTACTS AND LOCATIONS:
Overall Officials: Rong Zheng, MD, Principal Investigator — National Cancer Center/Cancer Hospital,Chinese Academy of Medical Sciences and PUMC
Locations (1):
- National Cancer Center/Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Chaoyang, China

IPD SHARING:
Plan to Share IPD: No